CLINICAL TRIAL: NCT01301040
Title: Early Detection of Chemotherapy Induced Cardiac Damage in Elderly Patients With Early Breast Cancer: a Randomized Phase II Trial Comparing (Neo) Adjuvant Epirubicin-cyclophosphamide (EC) Versus Docetaxel (Taxotere)-Cyclophosphamide (TC.)
Brief Title: Early Cardiac Toxicity of Adjuvant CT in Elderly BC.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Jules Bordet Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB 11-01; 2011-000562-35 (EudraCT Number)
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer
Keywords: breast cancer, elderly, early cardiac toxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epirubicin/Cyclophosphamide (Active Comparator): Treatment arm 1: EC - epirubicin (100mg/m2 IV) and cyclophosphamide (600mg/m2 IV) every 3 weeks for 4 cycles
  Interventions: Drug: epirubicin, cyclophosphamide, docetaxel
- docetaxel/cyclophosphamide (Active Comparator): Treatment Arm 2: TC - docetaxel (Taxotere) (75mg/m2 IV) and cyclophosphamide (600mg/m2 IV) every 3 weeks for 4 cycles.
  Interventions: Drug: epirubicin, cyclophosphamide, docetaxel

INTERVENTIONS:
Drug: epirubicin, cyclophosphamide, docetaxel — * Treatment arm 1: EC - epirubicin (100mg/m2 IV) and cyclophosphamide (600mg/m2 IV) every 3 weeks for 4 cycles.
  * Treatment Arm 2: TC - docetaxel (75mg/m2 IV) and cyclophosphamide (600mg/m2 IV) every 3 weeks for 4 cycles.
  Other Names: Docetaxel: Taxotere; Cyclophosphamide: Endoxan; Epirubicin: Epirubicin Teva

SUMMARY:
The primary objective is to evaluate the difference in cardiac strain rate evolution in elderly early BC patients treated with (neo) adjuvant anthracycline-based chemotherapy compared with a non-anthracycline regimen (Taxotere-cyclophosphamide) CT.

This study also will compare the serum biomarkers profile during and after the (neo) adjuvant CT in both treatment arms, assess whether MRI allows detecting earlier than standard echocardiography the signs of cardiotoxicity, during and after adjuvant (neo) CT, assess whether brain PET-CT allows detecting regional functional impairment in patients receiving CT, evaluate cognitive function before and after (neo) adjuvant CT in both treatment arms, evaluate distress and functional autonomy before and after (neo) adjuvant CT in both treatment arms, evaluate psychological state and burden of primary caregivers before and after (neo) adjuvant CT in both treatment arms, evaluate primary caregivers abilities to detect patients' distress and functional autonomy before and after (neo) adjuvant CT in both treatment arms, evaluate the short and long-term toxicity profile of the regimens, estimate the 10-year risk of relapse and/or death using the Adjuvant!Online tool, and estimate the Framingham risk score for Hard Coronary Heart Disease (10-year risk).

DETAILED DESCRIPTION:
Considering that both anthracycline-based and Taxotere-cyclophosphamide CT have established efficacy in the adjuvant treatment of elderly patients with early breast cancer, and the paucity of data for early cardiac toxicities with anthracycline-based adjuvant therapy compared to non-anthracycline regimen, this is the first randomized study to evaluate early cardiac signs based on doppler myocardial imaging (DMI). The results of this study could improve the monitoring of the cardiac function of elderly patients candidates to receive adjuvant chemotherapy for early breast cancer.

ELIGIBILITY:
1. Patient selection criteria

   * Female aged equal or more than 65 years.
   * Histological diagnosis of early BC for which the treating physician considers (neo) adjuvant chemotherapy to be beneficial. Recommended situations are:
   * Triple negative BC if pT > 1cm.
   * HER-2 positive BC if pT1 > 1cm; and trastuzumab will be given after study chemotherapy.
   * "Luminal B" cancers defined as ER+, PgR + or neg, Ki-67 ≥ 14%, and pT1 > 1cm.
   * "Luminal A" cancers (ER+, PgR+ and Ki-67 < 14%) will be considered only if ≥ 4 nodes.
   * Poor response to a preoperative endocrine therapy.
   * WHO performance status equal or less than 1.
   * Baseline LVEF equal or more than 50% measured by echocardiography.
   * Adequate organ function including:
   * neutrophils more or equal to 1.5 x 109/L.
   * platelets more or equal to100 x 109/L.
   * bilirubin < 1.25 x upper limit of normal (ULN) for the institution.
   * transaminases: AST < 2.5 x ULN , ALT < 2.5 x ULN and alkaline phosphatase ≤ 2.5 x ULN for the institution.
   * Estimated creatinine clearance > 30ml/min (using the Crockoft and Gault formula) (See Appendix E) .
   * No previous exposure to chemotherapy in this neoadjuvant or adjuvant setting.
   * No serious cardiac illness or medical conditions as judged by the investigator including, but not confined to:Symptomatic ventricular arrhythmias,Clinical and/or ECG evidence of myocardial infarction within the last 12 months,Coronary artery disease requiring medication,High-risk uncontrolled arrhythmias,Poorly controlled hypertension (e.g. systolic >180 mm Hg or diastolic >100 mm Hg).
   * Other concurrent serious diseases that may interfere with planned treatment including severe pulmonary conditions/illness.
   * No participation to other clinical trials involving therapeutic agents within the 6 weeks prior to the randomization.
   * No prior or concurrent diagnosis of cancer, except for adequately treated basocellular and squamous cell carcinoma of the skin or cervical uterine in situ tumor
   * Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
   * Signed written informed consent must be given according to ICH-GCP and national/local regulations, prior to any study specific screening procedures and randomization.
2. Caregiver selection criteria

   * to be identified by participating patients as their primary caregivers i.e the person who helps them the most to cope with cancer in their everyday life
   * to be at least eighteen years old
   * to be aware of the cancer diagnosis of the patients to be fit enough to complete the questionnaires
   * to be French speaking
   * to be free of any cognitive dysfunction.
   * to give their written informed consent as regards participation in the study.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The difference between cardiac strain rates measured at baseline and after 4 cycles of chemotherapy. | Before chemotherapy, after chemotherapy, at 6 months, one , two and 3 years from randomization.
  The primary null hypothesis is that the means are equal versus the alternative hypothesis that the means are different. We plan to perform the comparison using a two-sided Student's t-test with α=5%. The power of the study to detect the difference described below has been set at 90%.
  One hundred twenty patients candidate to receive neoadjuvant or adjuvant CT for early BC will be randomized 1:1 to receive either epirubicin-cyclophosphamide (EC) or docetaxel (Taxotere) -cyclophosphamide (TC) for 4 cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Lissandra Dal Lago, MD, Principal Investigator — Jules Bordet Institute; Evandro De Azambuja, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium